CLINICAL TRIAL: NCT03529916
Title: Endothelial Cell Gene Networks of CVD
Status: Withdrawn | Type: Observational
Why Stopped: No eligible participants were recruited
Sponsor: Tufts University (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Stefania lamon-Fava, Scientist I, Associate Professor, Tufts University
Other Study IDs: 12841
Record Dates: First submitted 2018-04-23; First posted 2018-05-18 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood will be obtained and subjected to isolation of circulating endothelial progenitor cells using pre-specified antibody micro-beads.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CVD subjects: CVD will be defined as >50% stenosis of one or more coronary arteries as assessed by coronary angiography.
  Interventions: Other: isolation of endothelial cells precursors in blood
- healthy controls: healthy controls defined as not having stenosis of coronary arteries as assessed by coronary angiography.
  Interventions: Other: isolation of endothelial cells precursors in blood

INTERVENTIONS:
Other: isolation of endothelial cells precursors in blood — Circulating endothelial precursor cells will be isolated and then cultured in vitro. RNA will be then isolated.

SUMMARY:
The objective of this study is to identify relevant signature gene networks of cardiovascular disease in endothelial cells derived from circulating endothelial progenitor cells of individuals with established cardiovascular disease (CVD).

DETAILED DESCRIPTION:
The investigators propose to enroll CVD and healthy subjects between 30 and 60 years of age, matched for age, gender, body mass index, and medication (statin and anti-hypertensive) use. Circulating endothelial progenitor cells will be isolated from blood and cultured in vitro to differentiate into endothelial cells.

ELIGIBILITY:
Inclusion Criteria for CVD subjects::

• >50% stenosis of one or more coronary arteries

Inclusion Criteria for Healthy subjects:

• absence of coronary artery stenosis

Exclusion Criteria for all subjects:

* type 2 diabetes mellitus
* chronic kidney disease,
* other chronic diseases
* dyslipidemia (fasting plasma LDL-C >160 mg/dL and triglyceride levels >150 mg/dL)

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Both CVD and healthy subjects
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2021-09-23 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Gene expression | 10 weeks
  Gene expression [ identify relevant signature gene networks of cardiovascular disease in endothelial cells]

CONTACTS AND LOCATIONS:
Overall Officials: Stefania Lamon-Fava, PhD, Principal Investigator — Tufts University
Locations (1):
- Tufts Medical Center - Cardiovascular Clinic, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No